CLINICAL TRIAL: NCT02653482
Title: Dapagliflozin Effect on Symptoms and Biomarkers in Patients With Heart Failure
Acronym: DEFINE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00032
Record Dates: First submitted 2016-01-04; First posted 2016-01-12 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Chronic Heart Failure With Reduced Systolic Function
Keywords: heart failure; dapagliflozin; Sodium-glucose co-transporter-2 (SGLT-2) inhibitors
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin 10 mg daily
  Interventions: Drug: Dapagliflozin
- Dapagliflozin matching placebo (Placebo Comparator): Dapagliflozin matching placebo 10 mg daily
  Interventions: Drug: Dapagliflozin matching placebo

INTERVENTIONS:
Drug: Dapagliflozin
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Dapagliflozin matching placebo
  Other Names: Placebo
  Arms: Dapagliflozin matching placebo

SUMMARY:
The primary purpose of this study is to evaluate the impact of dapagliflozin, as compared with placebo, on heart failure disease-specific biomarkers, symptoms, health status, and quality of life in patients with chronic heart failure with reduced systolic function.

DETAILED DESCRIPTION:
A 12-week randomized, double-blind, placebo-controlled trial to evaluate the effects of once-daily dapagliflozin 10 mg on heart failure disease-specific biomarkers (BNP and NTproBNP), symptoms, health status, and quality of life in patients with chronic heart failure with reduced systolic function.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of New York Heart Association (NYHA) Class II or Class III heart failure (left ventricular ejection fraction ≤40% due to either ischemic or non-ischemic etiology) with reduced systolic function for at least 16 weeks prior to enrollment
2. No change in diuretic management for at least 1 week prior to enrollment
3. Brain natriuretic peptide (BNP) ≥100 pg/mL and/or N-terminal pro b-type natriuretic peptide (NTproBNP) ≥ 400 pg/mL at enrollment

Exclusion Criteria:

1. History of type 1 diabetes
2. Estimated glomerular filtration rate (eGFR) < 30 at enrollment
3. Hospitalization for heart failure within the 30 days prior to enrollment
4. Admission for an acute coronary syndrome (ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, or unstable angina), percutaneous coronary intervention, or cardiac surgery within the 30 days prior to enrollment
5. Admission for cardiac resynchronization therapy (CRT) within 90 days prior to the screening visit
6. Planned cardiovascular revascularization (percutaneous intervention or surgical) or major cardiac surgery (coronary artery bypass grafting, valve replacement, ventricular assist device, cardiac transplantation, or any other surgery requiring thoracotomy) within the 90 days after enrollment
7. Patients who are volume depleted based upon physical examination at the time of screening or randomization

Ages: 19 Years to 119 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kosiborod, MD, Study Chair — Saint Luke's Mid America Heart Institute
Locations (25):
- United States (25):
  - Heart Group of the Eastern Shore, Fairhope, Alabama
  - University of Southern Califiornia, Los Angeles, California
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Emory University, Atlanta, Georgia
  - NorthShore University HealthSystem Research Institute, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - Advocate Health and Hospitals, Oakbrook Terrace, Illinois
  - University of Maryland, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Freeman Health System, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - New York University, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University, Durham, North Carolina
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nassif ME, Windsor SL, Tang F, Khariton Y, Husain M, Inzucchi SE, McGuire DK, Pitt B, Scirica BM, Austin B, Drazner MH, Fong MW, Givertz MM, Gordon RA, Jermyn R, Katz SD, Lamba S, Lanfear DE, LaRue SJ, Lindenfeld J, Malone M, Margulies K, Mentz RJ, Mutharasan RK, Pursley M, Umpierrez G, Kosiborod M. Dapagliflozin Effects on Biomarkers, Symptoms, and Functional Status in Patients With Heart Failure With Reduced Ejection Fraction: The DEFINE-HF Trial. Circulation. 2019 Oct 29;140(18):1463-1476. doi: 10.1161/CIRCULATIONAHA.119.042929. Epub 2019 Sep 16. PMID 31524498
- [Derived] Selvaraj S, Patel S, Sauer AJ, McGarrah RW, Jones P, Kwee LC, Windsor SL, Ilkayeva O, Muehlbauer MJ, Newgard CB, Borlaug BA, Kitzman DW, Shah SJ, Margulies KB, Husain M, Inzucchi SE, McGuire DK, Lanfear DE, Javaheri A, Umpierrez G, Mentz RJ, Sharma K, Kosiborod MN, Shah SH. Metabolic Effects of the SGLT2 Inhibitor Dapagliflozin in Heart Failure Across the Spectrum of Ejection Fraction. Circ Heart Fail. 2024 Nov;17(11):e011980. doi: 10.1161/CIRCHEARTFAILURE.124.011980. Epub 2024 Oct 18. PMID 39421941
- [Derived] Nassif ME, Windsor SL, Gosch K, Borlaug BA, Husain M, Inzucchi SE, Kitzman DW, McGuire DK, Pitt B, Scirica BM, Shah SJ, Umpierrez G, Austin BA, Lamba S, Khumri T, Sharma K, Kosiborod MN. Dapagliflozin Improves Heart Failure Symptoms and Physical Limitations Across the Full Range of Ejection Fraction: Pooled Patient-Level Analysis From DEFINE-HF and PRESERVED-HF Trials. Circ Heart Fail. 2023 Jul;16(7):e009837. doi: 10.1161/CIRCHEARTFAILURE.122.009837. Epub 2023 May 19. PMID 37203441
- [Derived] Selvaraj S, Fu Z, Jones P, Kwee LC, Windsor SL, Ilkayeva O, Newgard CB, Margulies KB, Husain M, Inzucchi SE, McGuire DK, Pitt B, Scirica BM, Lanfear DE, Nassif ME, Javaheri A, Mentz RJ, Kosiborod MN, Shah SH; DEFINE-HF Investigators. Metabolomic Profiling of the Effects of Dapagliflozin in Heart Failure With Reduced Ejection Fraction: DEFINE-HF. Circulation. 2022 Sep 13;146(11):808-818. doi: 10.1161/CIRCULATIONAHA.122.060402. Epub 2022 May 23. PMID 35603596
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: Drug information for dapagliflozin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0461432268&QV1=DAPAGLIFLOZIN

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: Dapagliflozin 10 mg daily
  Dapagliflozin
- Dapagliflozin Matching Placebo: Dapagliflozin matching placebo 10 mg daily
  Dapagliflozin matching placebo
Period: Overall Study
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Started | 131 | 132
Completed | 130 | 131
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo | Total
Number analyzed (Participants) | 131 | 132 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.0) | 60.4 (12.0) | 61.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 95 | 98 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 52 | 99
  White | 74 | 70 | 144
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 131 | 132 | 263
Duration of Heart Failure [Mean (Standard Deviation); unit: years] | 7.1 (5.8) | 7.2 (6.8) | 7.1 (6.3)
Previous Hospitalization for Heart Failure [Count of Participants; unit: Participants] | 101 | 108 | 209
Time since last hospitalization for heart failure [Mean (Standard Deviation); unit: years] | 1.4 (2.3) | 1.8 (3.1) | 1.6 (2.7)
Ejection fraction [Mean (Standard Deviation); unit: %] | 27.2 (8.0) | 25.7 (8.2) | 26.4 (8.1)
Ischemic heart disease [Count of Participants; unit: Participants] | 70 | 69 | 139
Type 2 diabetes mellitus [Count of Participants; unit: Participants] | 81 | 85 | 166
Atrial Fibrillation [Count of Participants; unit: Participants] | 57 | 49 | 106
Internal Cardiac Defibrillator (ICD) [Count of Participants; unit: Participants] | 88 | 75 | 163
Cardiac resynchronization therapy (CRT) [Count of Participants; unit: Participants] | 43 | 25 | 68
Angiotensin converting enzyme inhibitor (ACEI) / Angiotensin II receptor blocker (ARB) [Count of Participants; unit: Participants] | 76 | 80 | 156
Angiotensin receptor-neprilysin inhibitor (ARNI) [Count of Participants; unit: Participants] | 47 | 38 | 85
β-blockers [Count of Participants; unit: Participants] | 130 | 124 | 254
Hydralazine [Count of Participants; unit: Participants] | 19 | 26 | 45
Long-acting nitrates [Count of Participants; unit: Participants] | 17 | 22 | 39
Mineralocorticoid receptor agonist (MRA) [Count of Participants; unit: Participants] | 76 | 84 | 160
Loop diuretics [Count of Participants; unit: Participants] | 114 | 111 | 225
Digoxin [Count of Participants; unit: Participants] | 25 | 21 | 46
Lipid-lowering agents [Count of Participants; unit: Participants] | 107 | 104 | 211
Anticoagulant agent [Count of Participants; unit: Participants] | 58 | 42 | 100
Insulin - among patients with type 2 diabetes [Count of Participants; unit: Participants] | 42 | 45 | 87
Glucagon-like peptide-1 receptor agonist (GLP-1RA ) - among patients with type 2 diabetes [Count of Participants; unit: Participants] | 4 | 1 | 5
Dipeptidyl Pepdidase 4 (DPP4) inhibitor - among patients with type 2 diabetes [Count of Participants; unit: Participants] | 11 | 10 | 21
Sulfonylurea - among patients with type 2 diabetes [Count of Participants; unit: Participants] | 20 | 15 | 35
Metformin - among patients with type 2 diabetes [Count of Participants; unit: Participants] | 29 | 33 | 62
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 30.7 [27.3 to 35.9] | 30.6 [27.6 to 36.4] | 30.6 [27.5 to 36.3]
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 72.2 (12.4) | 71.8 (11.3) | 71.9 (12.3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 122.3 (20.1) | 124.8 (21.6) | 123.7 (20.2)
N-terminal pro B-type natriuretic peptide (NT-proBNP) [Median (Inter-Quartile Range); unit: pg/mL] | 1136 [668 to 2465] | 1136 [545 to 2049] | 1136 [615 to 2266]
Brain natriuretic peptide (BNP) [Median (Inter-Quartile Range); unit: pg/mL] | 288 [158 to 592] | 242 [138 to 542] | 269 [142 to 570]
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m2] | 66.9 (21.1) | 71.2 (23.1) | 69.1 (22.2)
Urine Albumin/Creatinine Ratio [Mean (Inter-Quartile Range); unit: mg/g] | 19.0 [7.0 to 87.0] | 25.0 [6.5 to 103.0] | 22.0 [7.0 to 96.0]
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 7.0 (1.8) | 7.3 (2.0) | 7.2 (1.9)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.5 (1.9) | 13.3 (1.7) | 13.4 (1.8)
New York Heart Association (NYHA) Class II [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina. A higher class means a worse functional condition.
  NYHA Class II indicates the patient has been classified as having slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 91 | 82 | 173
New York Heart Association (NYHA) Class III [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina. A higher class means a worse functional condition.
  NYHA Class III indicates the patient has been classified as having marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Participants | 40 | 50 | 90
Kansas City Cardiomyopathy Questionnaire - Overall Summary Score (KCCQ-OS) [Mean (Standard Deviation); unit: score on a scale] — The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status.
  score on a scale | 67.4 (22.0) | 67.0 (21.1) | 67.2 (21.5)
Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CS) [Mean (Standard Deviation); unit: score on a scale] — The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status.
  score on a scale | 70.8 (21.9) | 69.9 (21.4) | 70.3 (21.6)
6-minute walk distance [Median (Inter-Quartile Range); unit: meters] | 306 [243 to 368] | 305 [227 to 372] | 305 [229 to 369]

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Average of the 6- and 12-week Mean N-terminal Pro B-type Natriuretic Peptide (NTproBNP).
Description: Difference in the average of the 6- and 12-week mean N-terminal pro B-type natriuretic peptide (NTproBNP).
Time Frame: Average of Week 6 and Week 12
Population: The number of participants analyzed may differ from the overall number of participants analyzed due to missing data at certain timepoints for some participants.
Measure: Mean (95% Confidence Interval); unit: pg/dL
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
pg/dL | 1133 [1036 to 1238] | 1191 [1089 to 1304]

2. Primary Outcome: Percentage of Patients That Achieve a ≥ 5-point Increase in Heart Failure Disease Specific Quality of Life (Assessed Using Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS)) or a ≥ 20% Decrease in NTproBNP Over 12 Weeks
Description: A composite of the percentage of patients that achieved a meaningful improvement in health status (≥5-point increase in average of 6- and 12-week KCCQ-OS) or NT-proBNP (≥20% decrease in average of 6- and 12-week NT-proBNP).
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the KCCQ overall summary score, a small but clinically meaningful change is considered to be ≥ 5 points.
Time Frame: Average of Week 6 and Week 12
Population: as for outcome 1
Measure: Number; unit: % of participants
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
% of participants | 61.5 | 50.4

3. Secondary Outcome: Percentage of Patients With a ≥ 5-point Increase in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS)
Description: Percentage of patients with a ≥ 5-point increase in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) as measured at Week 6 and Week 12.
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the KCCQ overall summary score, a small but clinically meaningful change is considered to be ≥ 5 points.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
Participants
  Week 6 - Improvement in KCCQ-OS: number analyzed (Participants) | 126 | 128
  Week 6 - Improvement in KCCQ-OS | 59 | 46
  Week 12 - Improvement in KCCQ-OS: number analyzed (Participants) | 126 | 126
  Week 12 - Improvement in KCCQ-OS | 54 | 41

4. Secondary Outcome: Percentage of Patients With a ≥ 20% Decrease in N-terminal Pro B-type Natriuretic Peptide (NTproBNP)
Description: Percentage of patients with a ≥ 20% decrease in NTproBNP as measured at Week 6 and Week 12.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
Participants
  NTproBNP decrease ≥ 20 % at Week 6: number analyzed (Participants) | 125 | 126
  NTproBNP decrease ≥ 20 % at Week 6 | 43 | 42
  NTproBNP decrease ≥ 20 % at Week 12: number analyzed (Participants) | 125 | 126
  NTproBNP decrease ≥ 20 % at Week 12 | 55 | 37

5. Secondary Outcome: Percentage of Patients With a ≥ 5-point Increase in Kansas City Cardiomyopathy Questionnaire - Overall Summary Score (KCCQ-OS) and a ≥ 20% Decrease in N-terminal Pro B-type Natriuretic Peptide (NTproBNP)
Description: The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the KCCQ overall summary score, a small but clinically meaningful change is considered to be ≥ 5 points.
Time Frame: Average of Week 6 and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
Participants | 20 | 17

6. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) Over 12 Weeks.
Description: Change in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) over 12 weeks as measured at Week 6 and Week 12.The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the KCCQ overall summary score, a small but clinically meaningful change is considered to be ≥ 5 points.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
score on a scale
  KCCQ-OS - week 6: number analyzed (Participants) | 126 | 128
  KCCQ-OS - week 6 | 71.1 [68.7 to 73.5] | 70.1 [67.7 to 72.5]
  KCCQ-OS - week 12: number analyzed (Participants) | 126 | 126
  KCCQ-OS - week 12 | 72.6 [70.2 to 75.0] | 68.9 [66.5 to 71.4]

7. Secondary Outcome: Change in 6 Minute Walk Score Over 12 Weeks.
Description: Change in 6 minute walk score over 12 weeks as measured at Week 6 and Week 12. The 6 minute walk test measures the distance in meters that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
meters
  6-minute walk distance - 6 weeks: number analyzed (Participants) | 122 | 126
  6-minute walk distance - 6 weeks | 297.1 [285.1 to 309.6] | 289.6 [278.0 to 301.7]
  6-minute walk distance - 12 weeks: number analyzed (Participants) | 117 | 123
  6-minute walk distance - 12 weeks | 303.7 [291.2 to 316.7] | 301.3 [289.1 to 313.9]

8. Secondary Outcome: Change in Brain Natriuretic Peptide (BNP) Over 12 Weeks.
Description: Change in BNP over 12 weeks as measured at Week 6 and Week 12 as measured at Week 6 and Week 12.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
pg/mL
  BNP - week 6: number analyzed (Participants) | 124 | 127
  BNP - week 6 | 236 [212 to 263] | 265 [238 to 296]
  BNP - week 12: number analyzed (Participants) | 124 | 124
  BNP - week 12 | 228 [204 to 254] | 272 [243 to 303]

9. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) Over 12 Weeks.
Description: Change in HbA1c over 12 weeks as measured at Week 6 and Week 12.
Time Frame: Baseline to Week 6 and Week 12
Population: The number analyzed may differ from the overall number analyzed due to missing data at certain timepoints for some participants.
Measure: Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
percentage of glycated hemoglobin
  HbA1c - week 6: number analyzed (Participants) | 125 | 127
  HbA1c - week 6 | 6.9 [6.8 to 7.1] | 7.1 [7.0 to 7.2]
  HbA1c - week 12: number analyzed (Participants) | 125 | 126
  HbA1c - week 12 | 6.9 [6.8 to 7.1] | 7.1 [7.0 to 7.2]

10. Secondary Outcome: Change in Weight Over 12 Weeks
Description: Change in weight over 12 weeks as measured at Week 6 and Week 12.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
kg
  Weight - week 6: number analyzed (Participants) | 125 | 127
  Weight - week 6 | 96.0 [95.4 to 96.5] | 96.6 [96.0 to 97.1]
  Weight - week 12: number analyzed (Participants) | 126 | 128
  Weight - week 12 | 96.3 [95.7 to 96.8] | 96.6 [96.0 to 97.1]

11. Secondary Outcome: Change in Systolic Blood Pressure Over 12 Weeks
Description: Change in systolic blood pressure over 12 weeks as measured at Week 6 and Week 12.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
Number analyzed (Participants) | 130 | 129
mm Hg
  Systolic Blood Pressure - week 6: number analyzed (Participants) | 125 | 127
  Systolic Blood Pressure - week 6 | 119.2 [116.6 to 121.9] | 121.1 [118.5 to 122.4]
  Systolic Blood Pressure - week 12: number analyzed (Participants) | 126 | 128
  Systolic Blood Pressure - week 12 | 120.9 [118.2 to 123.5] | 119.8 [117.2 to 122.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 15 weeks. The adverse event collection period started at the time the patient signed consent at their Screening Visit, continued through a 12-week double-blind treatment period after randomization, and ended after completion of a 1-week follow-up period after completion of the double-blind treatment period.
Description: Serious Adverse Events, Drug Adverse Events, Adverse Events of Special Interest and Urgent Outpatient Heart Failure Visits were collected. A Drug Adverse Event is an adverse event which leads to premature and permanent discontinuation of study medication. Adverse Events of Special Interest include diabetic ketoacidosis, volume depletion (defined as hypotension, syncope, orthostatic hypotension or dehydration), severe hypoglycemic events and lower limb amputations.
Arm/Group | Dapagliflozin | Dapagliflozin Matching Placebo
All-Cause Mortality (participants affected / at risk) | 1/131 | 1/132
Serious Adverse Events (participants affected / at risk) | 32/131 | 31/132
Other Adverse Events (participants affected / at risk) | 19/131 | 18/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=131) | Dapagliflozin Matching Placebo (N=132)
Exacerbation of Heart Failure (Cardiac disorders) | 14 (26) | 14 (19)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
Acute Dyspnea (General disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (General disorders) | 1 (1) | 1 (1)
Acute Respiratory Distress (General disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atypical Chest Pain (General disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cachexia (General disorders) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Cerebrovascular Accident (General disorders) | 0 (0) | 2 (2)
Chest Pain (General disorders) | 1 (1) | 4 (6)
Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cocaine Abuse (General disorders) | 1 (1) | 0 (0)
Elevated Cardiac Enzymes (Cardiac disorders) | 0 (0) | 1 (1)
Epistaxis (General disorders) | 0 (0) | 1 (1)
Exacerbation of COPD (General disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gout (General disorders) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Hypertensive Urgency (General disorders) | 0 (0) | 1 (1)
ICD Implantation (Cardiac disorders) | 0 (0) | 3 (3)
ICD Shock due to Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Left Great Toe Infection (Infections and infestations) | 1 (1) | 0 (0)
Morbid Obesity - Remove Laparoscopic band (General disorders) | 0 (0) | 1 (1)
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non Intractable Headache (General disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pre-Renal Acute Kidney Injury (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock secondary to purulent skin infection from herpes zoster (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (General disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (General disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Volume Depletion (General disorders) | 2 (2) | 1 (1)
Worsening Coronary Artery Disease (Cardiac disorders) | 2 (2) | 1 (1)
Worsening Peripheral Artery Disease (General disorders) | 1 (1) | 0 (0)
Oliguric Acute Kidney Injury on CKD III (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=131) | Dapagliflozin Matching Placebo (N=132)
Urgent Heart Failure Visit (Cardiac disorders) | 3 (4) | 7 (12)
Volume Depletion (General disorders) | 10 (12) | 7 (7)
Severe Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1)
Hypotension (General disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (General disorders) | 1 (1) | 0 (0)
Vaginal Discharge (General disorders) | 1 (1) | 0 (0)
Bullae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Atypical Chest Pain (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-11-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT02653482/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT02653482/SAP_001.pdf